CLINICAL TRIAL: NCT00720993
Title: Altered Gene Expression in Colorectal "Smears" of Individuals With Colon Cancer
Brief Title: Colorectal Cancer Screening Validation Study
Acronym: CRC screening
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: IntelliGeneScan, Inc. (Industry)
Collaborators: BiotechNiks / Molecular Medicine Research Institute (Unknown)
Responsible Party: Lothar Wieczorek, PhD, Clinical and Regulatory Consultant, IntelliGeneScan, Inc.
Other Study IDs: IGS-08-001
Record Dates: First submitted 2008-07-21; First posted 2008-07-23 (Estimated); Last update posted 2009-04-23 (Estimated); Status verified 2009-02

CONDITIONS: Colorectal Cancer Screening
Keywords: Colorectal cancer screening; Gene expression; RTPCR

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Rectal smears ("cytology brush") samples and RNA recovered from such materials.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Control group - patients scheduled for routine colonoscopy procedures with no self or family history or other GI conditions.
- 2: Case group - patients with confirmed colorectal carcinoma scheduled for surgery or observed during routine colonoscopy screening.

SUMMARY:
The purpose of this study is to evaluate the gene expression patterns from colorectal mucosal cells collected through the use of a standard anoscope and cytology brush. Patients will include those scheduled for routine colonoscopy procedures and those with confirmed colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* willing to provide informed consent
* greater than or equal to 50 years of age
* patient is scheduled for routine colonoscopy procedure or colorectal cancer surgery
* subject is willing to provide colorectal mucosal sample for gene expression testing

Exclusion Criteria:

* recent radiation or treatment for gynecologic, prostate or rectal cancer
* recent surgery for anal rectal disease
* polys, family or self history of cancer (control group only)
* GI disease
* any mucosal disease or systemic condition that may confound the scientific interpretation of the gene expression results

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing routine colonoscopy screening or patients scheduled for colorectal cancer surgery.
Sampling Method: Probability Sample
Enrollment: 165 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-05 (Estimated); Study Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
- To select a threshold for Mahalanobis distance to determine the best operating characteristics (sensitivity and specificity) in subjects with cancer and subjects without cancer. - To explore other empirical metrics based on previous exploratory data | Mai 2009

SECONDARY OUTCOMES:
- To obtain data to estimate sensitivity, specificity, and the ROC curve for a test based on M-distance. - To determine the variability of sensitivity and specificity estimates | Mai 2009

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States